CLINICAL TRIAL: NCT06154265
Title: Default vs As-Needed Intraoperative Transesophageal Echocardiography (TEE) in Low-Risk Isolated Coronary Artery Bypass Graft (CABG) Surgery: A Randomized Controlled Trial
Brief Title: Intraoperative Echocardiography in Low-Risk CABG Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 853364
Record Dates: First submitted 2023-11-13; First posted 2023-12-04 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Heart Diseases; Coronary Artery Disease; Chest Pain; Stenosis Coronary; STEMI
Keywords: Heart; Chest Pain; Artery; Stenosis; TEE; CABG; Bypass
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease; Chest Pain; Coronary Stenosis; ST Elevation Myocardial Infarction; Constriction, Pathologic | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Intervention Model Description: (1) Default TEE: Where the TEE probe is placed after going under general anesthesia and a breathing tube is placed. TEE issued to take pictures of your heart before and after the CABG surgery. The TEE probe will remain in place throughout the surgery. (2) As-Needed TEE: Where the TEE probe is placed only in situations where a surgeon requires information that can only be obtained by ultrasound imaging of the heart.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Default TEE (Active Comparator): The TEE probe is placed after going under general anesthesia and a breathing tube is placed. TEE issued to take pictures of the heart before and after a CABG surgery. If randomized to this group, the TEE probe will remain in place throughout the surgery.
  Interventions: Device: TEE probe
- As-needed TEE (Other): The TEE probe is placed only in situations where a surgeon requires information that can only be obtained by ultrasound imaging of the heart.
  Interventions: Device: TEE probe

INTERVENTIONS:
Device: TEE probe — Transesophageal echocardiography, ultrasound probe
  Other Names: Philips transesophageal echocardiography (TEE), ultrasound probe

SUMMARY:
This goal of this study is to better understand when and where intraoperative transesophageal echocardiography (TEE) should (or should not) be used during coronary artery bypass graft (CABG) surgeries.

DETAILED DESCRIPTION:
This trial will look at benefits and harms to two different treatments strategies in order to improve clinical outcomes. Intraoperative TEE is an ultrasound-based, imaging device that uses sound valves to look at the heart continuously during a heart surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo isolated CABG surgery at a hospital within the UPenn Health System
2. Age ≥18 years
3. Ejection fraction ≥50%
4. Transthoracic echocardiography within one year of scheduled surgery date
5. Left heart catheterization within one year of scheduled surgery date
6. English language fluency or facilitated via language interpreter
7. Able to provide informed consent either in English or via a language interpreter
8. Willing to comply with all study procedures

Exclusion Criteria:

1. Documented valve (aortic, mitral, tricuspid, or pulmonic) disease (stenosis or regurgitation) moderate or greater.
2. Any CABG surgery with either "possible" or "definite" aortic intervention listed as a planned part of the procedure. plan for either definite or possible surgical intervention.
3. Any CABG surgery with either "possible" or "definite" valve repair/replacement listed as a planned part of the procedure.
4. Having undergone any previous cardiac surgeries (i.e. scheduled with a "REDO" modifier).
5. Proximal/critical left main coronary disease (e.g. greater than or equal to 90% stenosis).
6. Preexisting anomalous coronary arteries
7. Preexisting end-stage renal disease on hemodialysis
8. Preexisting chronic kidney disease (CKD) stage 3, 4, or 5
9. Stroke with residual focal neurological deficit(s) within 90 days of surgery
10. Any of the following presurgical, mechanical circulatory support devices:

    1. Intraaortic balloon pump
    2. Percutaneous right ventricular assist device (RVAD)
    3. Impella
    4. Extracorporeal membrane oxygenation (ECMO)
11. Absolute contraindication to echocardiography defined as one or more of the following documented conditions:

    1. Esophagectomy
    2. Esophagogastrectomy
    3. Esophageal trauma
12. Any of these three relative contraindication to TEE:

    1. Esophageal varies
    2. Gastric bypass surgery
    3. Descending thoracic aortic aneurysm
13. Severe pulmonary hypertension defined as:

    1. Pulmonary arterial pressure ≥60 mmHg
    2. Pulmonary vascular resistance (PVR) ≥3 Woods Units
14. Hemodynamic instability after induction and following placement of an endotracheal tube will be defined as one or more of the following events or scenarios:

    1. Placement of an intraaortic balloon pump (IABP)
    2. Initiation of venoarterial extracorporeal membrane oxygenation (VAECMO)
    3. Placement of a right or left percutaneous mechanical circulatory support device
    4. Initiation of epinephrine infusion at a dose ≥ 6 mcg/min for a duration ≥5 minutes
    5. Initiation of norepinephrine at a dose ≥8 mcg/min for a duration ≥ minutes
    6. Initiation of phenylephrine infusion at a dose ≥100 mcg/min for a duration ≥ minutes
    7. Initiation of vasopressin infusion at a dose ≥0.04 units/min for a duration ≥ minutes

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Objectives | 24 months
  1. Recruitment feasibility assessment as measured by an absolute recruitment rate. Absolute recruitment rate is defined as the number of successfully enrolled participants divided by the total number of screened participants.
  2. Assess intervention fidelity by calculating the rate of TEE performed among participants randomized to the as-needed TEE trial arm.

SECONDARY OUTCOMES:
Secondary Objectives | 24 month
  1. Evidence of clinically-significant gastroesophageal dysfunction during hospitalization - either by patient-reported symptoms or by the presence of testing for swallowing difficulty, dysfunction, or upper endoscopy diagnostic procedures.
  2. Evidence of end-organ dysfunction based on clinical notes (e.g. "transaminitis," "acute kidney/renal injury"), and/or laboratory-based evidence of (e.g. liver function tests [LFTs], serum creatinine [Cr], lactate, etc.).
  3. Incidence of in-hospital, post-surgical, cardiovascular re-intervention (e.g. return to the operating room for any reason, unplanned or emergency cardiac catheterization post-surgery, or placement on venoarterial extracorporeal membrane oxygenation [VAECMO]).
  4. Incidence of all-cause in-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Emily MacKay, DO, MS, Principal Investigator — University of Pennsylvania, Penn Medicine
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States